CLINICAL TRIAL: NCT05283967
Title: Urine Colorimetry for Tuberculosis Pharmacokinetics Evaluation in Children and Adults
Acronym: PEE-TB
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Rutgers, The State University of New Jersey (Other); University of Florida (Other)
Responsible Party: Principal Investigator, Scott Heysell, MD, Associate Professor of Medicine, Infectious Diseases and International Health, University of Virginia
Other Study IDs: 20944
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adults and children, U.S.: A prospective, observational study of the pharmacokinetics of first-line anti-TB drugs (isoniazid, rifampin, and pyrazinamide) among TB patients (i.e. patients with active TB disease) will be conducted.
  Interventions: Diagnostic Test: urine colorimetric assay
- Tanzanian children: A prospective, observational study of the pharmacokinetics of first-line anti-TB drugs (isoniazid, rifampin, and pyrazinamide) among TB patients (i.e. patients with active TB disease) will be conducted.
  Interventions: Diagnostic Test: urine colorimetric assay

INTERVENTIONS:
Diagnostic Test: urine colorimetric assay — Colorimetric assays will be performed for urine drug concentrations of rifampin, isoniazid and pyrazinamide from urine collected throughout one dosing interval. Assay results will experimental only and not used to change patient care.

SUMMARY:
The purpose of the study is to generate receiver-operating-characteristic (ROC) curves for urine colorimetry to identify tuberculosis (TB) patients (children and adults) with low drug anti-TB drug exposures, which will define the diagnostic accuracy. The central hypothesis is that urine colorimetry will successfully identify patients with low anti-TB serum drug levels, and do so with diagnostic characteristics similar to other widely used tests in TB management.

DETAILED DESCRIPTION:
TB remains a leading infectious disease cause-of-death worldwide, with an estimated 1.5 million TB deaths each year. There is wide variability in absorption and metabolism of the anti-TB drugs, and low drug concentrations in blood are associated with inferior TB treatment outcomes, including treatment failure, relapse, and the emergence of drug-resistant infections. According to the most recent CDC/ATS/IDSA guidelines for TB treatment, therapeutic drug monitoring should be routinely considered for use among patients in high-risk groups, including adults with co-morbid type 2 diabetes mellitus (DM) and children. However, therapeutic drug monitoring requires sophisticated laboratory techniques unavailable for millions of patients receiving TB therapy in resource-limited settings where the vast majority of TB cases are treated. A new approach to measuring anti-TB drug exposures, based on technology easily adapted to resource-limited settings, is vitally needed and would be in line the World Health Organization's goal of the optimization of anti-TB drug regimens as a key component of the End TB Strategy.

A simple, inexpensive test to identify pediatric and adult TB patients with low drug exposures, available at the point-of-care at the time of the patient encounter, would support clinical decision-making. The performance of therapeutic drug monitoring requires specialty laboratory capabilities, such as high-performance liquid chromatography or gas chromatography. Technical expertise is also required to collect, process, and ship samples to the specialty laboratory. In many high-burden settings, the complexity and cost of these laboratory methods preclude the use of therapeutic drug monitoring in the clinical care of tuberculosis patients. These complexities also foster a dependence of TB endemic sites on laboratories in resource-rich environments. Consequently, patients with inadequate drug exposures cannot be identified early in anti-TB therapy, at the critical time when dosing adjustments could be expected to improve treatment outcomes.

Urine colorimetry provides a low-technology approach for measuring anti-TB drug exposures, suitable for point-of-care testing. Colorimetry is the measurement of intensity of signal at a specific wavelength in the visible region of the spectrum. Urine colorimetry was evaluated as a method to assess the relative bioavailability of different fixed-dose combinations of anti-TB drugs administered to healthy volunteers. The study is based on the scientific premise that more detailed anti-TB drug exposure information can be obtained from urine sampling during TB treatment, not only to determine the presence or absence of drugs or metabolites, but to determine whether the presence of drugs or metabolites has surpassed a critical exposure threshold, informing drug dosing decision-making at the point-of-care. Potential advantages of urine colorimetric methods include a non-invasive sampling approach, improved patient acceptability, and the low cost and stability of chemical reagents. Colorimetry is particularly suited for point-of-care diagnostics, possibly with battery-operated or smartphone-based tools. With a simple diagnostic test available at the point-of-care, with results provided at the time of the clinical encounter, the TB clinician will be able to adjust drug doses and optimize regimens.

ELIGIBILITY:
Inclusion Criteria:

Patients of male and female sex meeting all of these criteria:

* Those 4 years and older;
* Diagnosed with active TB and initiation of combination anti-TB therapy with isoniazid, rifampin, and pyrazinamide, with or without DM;
* Able to provide informed consent and assent for those 7-17 years old.

Exclusion Criteria:

* Anuric (i.e. not capable of producing urine due to chronic renal disease);
* Pregnancy or breastfeeding;
* Prisoners

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study personnel will review the daily clinic rosters at each enrollment site to identify patients with TB who have initiated or are planning to initiate first-line anti-TB therapy with a regimen that includes isoniazid, rifampin, and pyrazinamide.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Urine Cmax | Day 1
  Urine peak concentration (Cmax) of rifampin as determined by urine colorimetry
Urine rifampin AUC | Day 1
  Urine total rifampin area under the concentration time curve (AUC) as determined by urine colorimetry
Urine isoniazid Cmax | Day 1
  Urine peak concentration (Cmax) of isoniazid as determined by urine colorimetry
Urine isoniazid AUC | Day 1
  Urine total isoniazid area under the concentration time curve as determined by urine colorimetry
Urine pyrazinamide Cmax | Day 1
  Urine peak concentration (Cmax) of pyrazinamide as determined by urine colorimetry
Urine pyrazinamide AUC | Day 1
  Urine total pyrazinamide area under the concentration time curve as determined by urine colorimetry

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rutgers, The State University of New Jersey, Newark, New Jersey
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
All study participant data will be maintained in a de-identified dataset. At study conclusion, investigators will determined plan for IPD sharing.

REFERENCES:
- [Background] Szipszky C, Van Aartsen D, Criddle S, Rao P, Zentner I, Justine M, Mduma E, Mpagama S, Al-Shaer MH, Peloquin C, Thomas TA, Vinnard C, Heysell SK. Determination of Rifampin Concentrations by Urine Colorimetry and Mobile Phone Readout for Personalized Dosing in Tuberculosis Treatment. J Pediatric Infect Dis Soc. 2021 Mar 26;10(2):104-111. doi: 10.1093/jpids/piaa024. PMID 32170944
- [Background] Zentner I, Modongo C, Zetola NM, Pasipanodya JG, Srivastava S, Heysell SK, Mpagama S, Schlect HP, Gumbo T, Bisson GP, Vinnard C. Urine colorimetry for therapeutic drug monitoring of pyrazinamide during tuberculosis treatment. Int J Infect Dis. 2018 Mar;68:18-23. doi: 10.1016/j.ijid.2017.12.017. Epub 2017 Dec 15. PMID 29253711
- [Derived] Petros de Guex K, Augustino D, Mejan P, Gadiye R, Massong C, Lukumay S, Msoka P, Sariko M, Kimathi D, Vinnard C, Xie Y, Mmbaga B, Pfaeffle H, Geba M, Heysell SK, Mduma E, Thomas TA. Roadblocks and resilience: A qualitative study of the impact of pediatric tuberculosis on Tanzanian households and solutions from caregivers. Glob Public Health. 2023 Jan;18(1):2196569. doi: 10.1080/17441692.2023.2196569. PMID 37021699